CLINICAL TRIAL: NCT05165173
Title: Almond Milk With Vitamin D: Impact on Vitamin D Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB202102986; OCR41655 (Other: UF OnCore)
Record Dates: First submitted 2021-12-17; First posted 2021-12-21 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Renal Insufficiency, Chronic; Kidney Failure, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: randomized comparator-controlled trial
Who Masked: Participant, Investigator
Masking Description: Participants will receive a coded sample that either contains 4000 IUs microparticles of vitamin D or 4000 IUs nanoparticles of vitamin D
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Based on estimated glomerular filtration rate (eGFR) and vitamin D levels, participants will be placed into the nanoparticle group.
  Interventions: Dietary Supplement: NanoD4CKD
- Comparator (Active Comparator): Based on the estimated glomerular filtration rate (eGFR) and vitamin D levels, participants will be placed into the microparticle group.
  Interventions: Dietary Supplement: MicroD4CKD

INTERVENTIONS:
Dietary Supplement: NanoD4CKD — Participants will receive a 7-day supply of the 4-ounce almond milk mixed with 4000 IUs of nanoparticles of D3 and instructed to consume it in the morning with a meal.
  Arms: Intervention
Dietary Supplement: MicroD4CKD — Participants will receive a 7-day supply of the 4-ounce almond milk mixed with 4000 IUs of microparticles of D3 and instructed to consume it in the morning with a meal.
  Arms: Comparator

SUMMARY:
The overall goal is to enhance vitamin D status in a safe and effective manner. A 3-week randomized comparator-controlled trial among a cohort of adults with CKD (stages 3-5) (n=24) will test the main objective: Evaluate the bioefficacy of D3 in micro- and nanoparticles (4000IUs) in almond milk with the sub-objective of: Explore the effect of D3 in micro- and nanoparticles (4000IUs) in almond milk on inflammation markers CRP, TNF-α and IL-6.

ELIGIBILITY:
Inclusion Criteria:

* adults who have been diagnosed with CKD
* have no GI disorders or GI disturbances
* age 18 years or older
* no food allergies or dietary restrictions
* all with no contraindications to consuming anything by mouth as per their physician

Exclusion Criteria:

* no diagnosis of CKD
* GI disorders
* gastrointestinal disturbances
* under 18 years old
* food allergies to almonds
* Dietary restrictions as medically indicated
* trouble chewing/swallowing as confirmed by physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-11-18 (Actual); Study Completion 2023-11-18 (Actual)

PRIMARY OUTCOMES:
Vitamin D | 21 days
  baseline to end line in the concentration of serum 25(OH)D3 between and within the control and intervention groups.

SECONDARY OUTCOMES:
Calcium | 21 days
  baseline to end line in the concentration of serum calcium between and within the control and intervention groups.
PTH | 21 days
  baseline to end line in the concentration of serum PTH between and within the control and intervention groups.
parent vitamin D | 21 days
  baseline to end line in the concentration of serum parent vitamin D between and within the control and intervention groups.
IL-6 | 21 days
  baseline to end line in the concentration of serum IL-6 between and within the control and intervention groups.
C-reactive protein | 21 days
  baseline to end line in the concentration of C-reactive protein between and within the control and intervention groups.
TNF-alpha | 21 days
  baseline to end line in the concentration of serum TNF-alpha between and within the control and intervention groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Andrade, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No